CLINICAL TRIAL: NCT04061564
Title: Vagal Nerve Stimulation for Intestinal Barrier Dysfunction in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: QMERC2018/83
Record Dates: First submitted 2019-07-18; First posted 2019-08-20 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2019-07

CONDITIONS: Intestinal Barrier Dysfunction
MeSH Terms: interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Proof of concept randomised, placebo controlled, single blinded, cross over study
Who Masked: Participant
Masking Description: The use of the device in a location which will not stimulate the vagal nerve
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active transcutaneous vagal nerve stimulation (Active Comparator): The participant will be administered vagal nerve stimulation to each ear (20 minutes in total)
  Interventions: Device: Vagal nerve stimulation
- Sham transcutaneous vagal nerve stimulation (Sham Comparator): The participant will be administered sham stimulation to each ear (20 minutes in total)
  Interventions: Device: Vagal nerve stimulation

INTERVENTIONS:
Device: Vagal nerve stimulation — The participant will be administered electrical stimulation at a level specifically set to their comfort. This will be performed using a TENS machine device.

SUMMARY:
This is a proof of concept randomised placebo controlled crossover trial to evaluate the effect of transcutaneous vagal nerve stimulation on a stress model of increased intestinal permeability in healthy human subjects.

Intestinal permeability perturbation is a phenomenon which is being increasingly recognised as a contributing factor to a multitude of diseases - including inflammatory bowel disease (IBD) and irritable bowel syndrome (IBS). There are currently limited effective treatment methods known to improve this intestinal permeability perturbation and the use of vagal nerve stimulation would present itself as an inexpensive, non-invasive and non-pharmacological method of reversing this dysfunction. Vagal nerve stimulation efficacy in reversing stress related intestinal barrier dysfunction is available from proof of concept animal models.

This mechanistic project is an important first step in this field of research and will serve as a basis for further research into the role of vagal nerve stimulation in intestinal barrier dysfunction.

DETAILED DESCRIPTION:
Stress - a state which evokes a 'fight or flight' or sympathetic response from the human organism - has been implicated in the propagation of inflammation in patients with inflammatory bowel disease (IBD). Indeed, the risk of relapse in both Crohns disease (CD) and Ulcerative colitis (UC) increases in the presence of both acute and chronic stress. The mechanism proposed for this phenomenon includes the ability of stress to induce a breakdown in intestinal barrier function via mast cell- and corticotropin releasing hormone (CRH)-dependent pathways. This intestinal barrier perturbation has been demonstrated experimentally in humans using stress paradigms which could be equated to the relatively mild stressful events experienced in every-day life.

The autonomic nervous system (ANS) appears to be playing a crucial role in stress-induced changes in intestinal permeability. Multiple in vitro and in vivo murine model studies have confirmed that both acute and chronic stress (induced in a mouse by various stress paradigms such as restraint and water emersion) can promote increased intestinal permeability. The underlying mechanism seems to be via the disruption of tight junction proteins along the paracellular space of the intestinal epithelium. The disruption of tight junctions in these stress paradigm models are dependent on acetylcholine and CRH. This effect on intestinal permeability appears to recover within 4 days in murine models.

Similar changes have been described in human models of acute stress. Barclay and Turnberg first showed that intestinal absorption of salt and water was reduced in healthy participants in response to acute stress induced by a short-term stressor paradigm. In this study, they used dichotomous listening as the physiological stressor, whereby the participant is asked to listen to two types of different genres of music in each ear whilst they completed a mentally challenging task. These physiological absorption changes to the intestine's barrier function were found to be mediated by a cholinergic-dependent mechanism. The same authors later showed similar effects with the physical stress paradigm of cold-induced pain in healthy volunteers. Although actual intestinal permeability changes were not measured at the time, one likely mechanism of permeability changes related to these alterations in electrolyte flux is via the claudin-2 paracellular channel, which has since been described. The configuration of this channel is related to ionic flux across the intestinal epithelium and, therefore, would render the epithelium more permeable in times of electrolyte flux. In more recent studies utilising the same cold-pain paradigm, changes in intestinal permeability were paralleled by the release of products of mast cell degranulation, tryptase and histamine. Such changes in intestinal permeability induced by acute stress were mimicked by peripheral administration of CRH and could be reversed by the administration of mast cell stabilisers.

A key role for the parasympathetic nervous system in the perturbation of intestinal permeability by severe physiological stress was derived from the effects of vagal nerve stimulation in animal models. Stimulation of the cervical vagal nerve for 10 minutes prior to giving mice a severe burn protected them from intestinal barrier perturbation and increased intestinal glial fibrillary acidic protein (FGAP) expression, a marker of enteric nervous system glial activation, in vitro and in vivo.This effect was likely, at least in part, due to an α7 acetylcholine receptor dependent mechanism that was demonstrated in both cultured intestinal epithelial cells as well as in enteric glial cells. Further studies have since supported this protective effect of vagal nerve stimulation, suggesting a role for the preservation of the number of dendritic cells in the mesenteric lymph as another potential mechanism.Moreover, the protective effect on the epithelial lining seemed to be via a locally-induced mechanism on the intestine rather than being dependent on a splenic-mediated process as the protective effect held true in splenectomised mice. Stimulation of the parasympathetic nervous system via the vagal nerve therefore seems to play a protective role in modulation of the intestinal barrier function with experimental evidence hinting at its ability to reverse stress induced changes in intestinal permeability.

These results are of significant interest given that the last decade has seen a number of studies supporting the theory of intestinal barrier perturbation in the pathogenesis of IBD.Additionally, the detection of antibodies directed against microbial antigens (such as 'ASCA' - epitopes of Saccharomyces cerevisiae and Flagellin CBir1) are found in the serum of patients prior to the development of IBD - indicating a disruption of the intestinal barrier function prior to the onset of disease. Furthermore, a genetic predisposition to intestinal barrier perturbation is considered to be a predisposing factor in the development of IBD. Given that it seems that the ANS has a significant role to play in the maintenance of the intestinal barrier function, it would be reasonable to conclude that alterations within the ANS in a susceptible individual may, at least in part, be implicated the development and flares of IBD.

Several serological and urinary markers have been validated as useful tools in measuring intestinal permeability changes in vivo. These include lipopolysaccharide-binding protein (LBP), CD-14 and intestinal-type fatty acid-binding protein (I-FABP) in the serum, as well as an orally-administered dual sugar solution and its by-products in serum and urine. Soluble CD-14 and LBP are part of the LPS inflammatory signalling pathway, thus their levels in serum have been shown to be objective markers for systemic immune activation and damage to gut epithelium. I-FABP is an intracellular protein expressed in the epithelial cells of the mucosal layer of the small and large intestine tissue and is prone to leakage into the blood stream from the enterocytes when intestinal mucosal damage occurs. The oral dual sugar test uses lactulose and rhamnose that are differentially absorbed in the intestine and excreted in the urine. The ratio of lactulose to rhamnose in the urine and serum can be used as a measure of small intestinal permeability when the urine is collected for two hours post ingestion of the test solution.

The therapeutic effect of vagal nerve stimulation in intestinal barrier dysfunction is an important area of study as it could lead to a novel and in-expensive method of treatment of conditions associated with intestinal barrier perturbation. In humans, the auricular branch of the vagus nerve is located directly under the skin, making it a suitable target for transcutaneous stimulation. A transcutaneous electrical nerve stimulation (TENS) device is thus a suitable non-invasive tool for the investigation of transcutaneous vagal nerve stimulation (tVNS) for reduction of intestinal permeability in humans and has been used in a number of studies utilizing the technique of tVNS in our laboratory.

Corticotropin releasing hormone (CRH) is naturally secreted from the healthy human hypothalamus during periods of stress. Intravenously administered CRH possesses the advantage of having a short half-life and is routinely clinically utilised in the diagnosis of Cushing's syndrome. Recent evidence has shown that injecting CRH intravenously reliably and significantly increases intestinal permeability in healthy volunteers with no significant adverse effects.This model will be used to induce increased intestinal permeability in healthy human volunteers in order to test the hypothesis that pre-treatment with vagal nerve stimulation can reduce the degree of intestinal permeability induced by CRH.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between the ages of 18 - 65
* Participants who are able to give informed consent
* Volunteers should be able to attend the Wingate institute on 2 occasions

Exclusion Criteria:

Inclusion criteria:

* Healthy males and females between the ages of 18 - 65
* Participants who are able to give informed consent
* Volunteers should be able to attend the Wingate institute on 2 occasions

Exclusion Criteria

* Inclusion criteria not met
* Past medical history of diabetes (type 1 or 2)
* Past medical history of inflammatory bowel disease, Coeliac disease, a diagnosis of irritable bowel syndrome or significant gastrointestinal symptoms not otherwise medically diagnosed
* Patients actively taking non-steroidal anti-inflammatory medications (NSAIDs) or corticosteroids
* Probiotic or antibiotic intake over the past 3 months
* Pregnant or breast feeding participants
* Participants with known or suspected disorders of the hypothalamo-pituatory axis
* Participants with a history of anaphylaxis
* Chronic disease or any regular medication intake not already specified above; in particular:
* Participants with known or suspected severe cardiac disease (e.g., symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure (CHF);
* Participants with clinically significant abnormal screening 3 lead Electrocardiogram (ECG) e.g. second and third degree heart block, prolonged QT interval, atrial fibrillation, atrial flutter, history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction);
* Participants who are implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, cochlear implant, sphenopalatine ganglion stimulator or occipital nerve stimulator).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
The effect of vagal nerve stimulation on corticotropin releasing hormone induced intestinal barrier dysfunction | 2 months
  Blood (Intestinal fatty acid binding protein, CD14, Lipopolysaccaride binding protein, dual sugar test result) and urine analyses (the dual sugar test) will be used to determine the intestinal barrier function before and after vagal nerve stimulation. Stress induced intestinal barrier dysfunction will be reproduced with the administration of corticotropin releasing hormone. Intestinal fatty acid binding protein, CD14, Lipopolysaccaride binding protein will be measured quantitatively using the enzyme-linked immunosorbent assay and results will be presented in microgram/litre
  . Serum and urine sugar concentrations will be measured using high performance liquid chromatography. Results will be presented as a ratio between the monosaccharide and di-saccharide sugar concentrations (i.e. lactulose to rhamnose and lactulose to mannitol ratios).

SECONDARY OUTCOMES:
The effect of vagal nerve stimulation on autonomic parameter - mean root square difference of RR intervals | 2 months
  Participants' autonomic parameters will be monitored during, before and after vagal nerve stimulation. The mean root square difference of RR intervals will be calculated using a mathematical equation which utilises the time difference between the R-R interval (in seconds) on electrocardiographic monitoring. The mean root square difference will be reported in milliseconds.
  Comparisons of these parameters will then be made between the active and sham interventions.
The effect of vagal nerve stimulation on autonomic parameter - low frequency to high frequency ratio of RR intervals | 2 months
  Participants' autonomic parameters will be monitored during, before and after vagal nerve stimulation. Low frequency to high frequency ratio of the RR intervals will be calculated using a mathematical equation which utilises the time difference between the R-R interval (in seconds) on electrocardiographic monitoring. Low frequency to high frequency ratio will be reported as a 'ratio' (no units).
  Comparisons of these parameters will then be made between the active and sham interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- The Wigate Institute, Barts and the London School of Medicine and Dentistry, London, United Kingdom